CLINICAL TRIAL: NCT00003956
Title: A Phase I Study of Continuous Oral Administration of SCH 66336 and 5-Fluorouracil/Leucovorin (5FU/LV) in Patients With Advanced Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067155; MSKCC-99020; SPRI-C98-564-01; NCI-G99-1540
Record Dates: First submitted 1999-11-01; First posted 2004-09-14 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2009-12

CONDITIONS: Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; unspecified adult solid tumor, protocol specific; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Fluorouracil; Leucovorin; lonafarnib

INTERVENTIONS:
Drug: fluorouracil
Drug: leucovorin calcium
Drug: lonafarnib

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase I trial to study the effectiveness of SCH 66336, fluorouracil, and leucovorin in treating patients who have advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety, tolerability, maximum tolerated dose, and dose limiting toxicity of oral SCH 66336 with fluorouracil and leucovorin calcium in patients with advanced malignancy. II. Assess the multiple dose pharmacokinetics of oral SCH 66336 when administered with fluorouracil and leucovorin calcium. III. Assess the pharmacokinetics of fluorouracil when administered with oral SCH 66336. IV. Assess antitumor activity of oral SCH 66336 with fluorouracil and leucovorin calcium in these patients.

OUTLINE: This is a dose escalation study of SCH 66336. Patients receive oral SCH 66336 twice daily for 56 days. Patients receive leucovorin calcium IV over 1-2 minutes immediately followed by fluorouracil IV over 1-2 minutes on days 1, 8, 15, 22, 29, and 36. Courses repeat every 56 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of SCH 66336. The maximum tolerated dose is defined as the dose at which no more than 1 of 6 patients experiences dose limiting toxicity (DLT) during course 1, with at least 2 patients experiencing DLT at the next higher level.

PROJECTED ACCRUAL: Approximately 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven malignancy for which no curative therapy exists At least 1 bidimensionally measurable lesion No acute or chronic leukemia or multiple myeloma No active CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG-WHO 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count greater than 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9.0 g/dL Hepatic: Bilirubin no greater than 2.0 mg/dL SGOT or SGPT no greater than 3 times upper limit of normal (ULN) (5 times ULN if elevations due to liver metastasis) Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No prior or concurrent QTc interval prolongation greater than 500 m/sec, unless approved by cardiology consult prior to study Other: No malabsorption syndrome due to surgery, prior disease, or other unknown reason No frequent vomiting or other medical condition that could interfere with oral medicine intake (e.g., partial bowel obstruction, external biliary diversion) No concurrent nonmalignant systemic disease making patient a poor risk for study No active uncontrolled infection Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior biologic therapy and recovered No prior allogeneic, syngeneic, or autologous bone marrow transplantation No prior peripheral blood stem cell transplantation No concurrent biologic therapy Chemotherapy: No more than 2 prior chemotherapy regimens At least 4 weeks since prior chemotherapy (6 weeks since mitomycin or nitrosoureas) and recovered No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy and recovered No prior wide field radiation (radiotherapy to at least 25% of bone marrow, including pelvic irradiation) No concurrent radiotherapy Surgery: Prior major gastrointestinal surgery allowed if recovered Other: At least 4 weeks since other prior investigational therapy and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 1999-04; Primary Completion 2001-01 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard B. Saltz, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States